CLINICAL TRIAL: NCT06592599
Title: A Safety, Feasibility and Efficacy Study of Gemcitabine Plus Docetaxel Plus Toripalimab (GDT) Induction as Part of a Curative Sequential Chemoradiation for Patients With Locoregional EBV Associated Nasopharyngeal Carcinoma (NPC)
Brief Title: Gemcitabine + Docetaxel + Toripalimab Induction in Epstein-Barr Virus (EBV) Associated Nasopharyngeal Carcinoma(NPC)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-75587; NCI-2025-00939 (Registry Identifier: National Cancer Institute Clinical Trials Reporting Program)
Record Dates: First submitted 2024-09-09; First posted 2024-09-19 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Nasopharyngeal Carcinoma
Keywords: gemcitabine; docetaxel; toripalimab
MeSH Terms: conditions — Nasopharyngeal Carcinoma | interventions — toripalimab

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Gemcitabine, Docetaxel and Capecitabine (Experimental): Patients will receive three q 21-day cycles of gemcitabine 1000 mg/m2 plus docetaxel 75 mg/m2 plus toripalimab 240 mg, followed by radiation to 70 Gy plus concurrent weekly cisplatin, 40 mg/m2 up to 7 doses, followed by adjuvant capecitabine 650 mg/m2 BID for one year plus toripalimab 240 mg q 21 days for 9 doses.
  Interventions: Drug: Toripalimab; Radiation: Concurrent Chemoradiation and Adjuvant treatment following Chemoradiation

INTERVENTIONS:
Drug: Toripalimab — Toripalimab will be administered 240 mg intravenously every three weeks in combination with the induction chemotherapy regimen for 3 cycles, and for 9 cycles as adjuvant treatment following radiation as specified in the overall sequential treatment plan.
Radiation: Concurrent Chemoradiation and Adjuvant treatment following Chemoradiation — Radiation treatment will be initiated 3-6 weeks following day 1 of the last induction cycle using institutional standards of care and support as follows:
  Intensity modulated radiotherapy, 70 Gy in 33 fractions M-F once daily plus cisplatin 40 mg/m2 IV weekly for up to 7 doses.
  Following the completion of concurrent chemoradiation, capecitabine will be administered using institutional standards of care as follows:
  Capecitabine 650 mg/m2 PO BID x 12 months beginning 12 to 16 weeks following the end of radiation treatment. Dose reductions and discontinuance of capecitabine will be according to the standard of care applied at the treating institution.
  Adjuvant Toripalimab 240 mg IV q 21d x 9 maximum doses will be initiated concurrently with the initiation of adjuvant capecitabine, beginning 12-16 weeks following the end of radiation.

SUMMARY:
The purpose of the research is to test the safety and efficacy of the investigational drug in human subjects with cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Eligible disease(s) / stage(s): Locoregionally advanced EBV positive NPC (T3-4, any N OR any T, N1-3. No M1) per AJCC v 8
2. Prior therapy: None for NPC permitted
3. Life expectancy: 3 months at least
4. Contraception requirements: Women of childbearing potential and male participants who are sexually active must agree to use a medically effective means of birth control during treatment with toripalimab and for 4 months after the last dose.
5. ECOG Performance Status of 0,1, or 2
6. Age: At least 18 years old.

   CBC/differential obtained within 21 days prior to day 1 of treatment, with adequate bone marrow function defined as follows:
7. Absolute neutrophil count (ANC) ≥ 1,500 cells/mm3
8. Platelets ≥ 100,000 cells/mm3;
9. Hemoglobin ≥ 8.0 g/dl (Note: The use of transfusion or other intervention to achieve Hgb ≥ 8.0 g/dl is acceptable.);

   Adequate hepatic function within 21 days prior to day 1 of treatment, defined as follows:
10. Total bilirubin ≤ 1.5 x institutional ULN;
11. AST and ALT ≤ 1.5 x institutional ULN;

    Adequate renal function within 21 days prior to day 1 of treatment, defined as follows:
12. Serum creatinine ≤ 1.5 mg/dl or calculated or measured creatinine clearance (CC) ≥ 50 ml/min
13. Negative serum pregnancy test within 14 days prior to day 1 of treatment for women of childbearing potential
14. Ability to understand and the willingness to personally sign the written IRB approved informed consent document.

Exclusion Criteria:

1. Prior systemic anticancer treatment for NPC
2. Prior radiation to head and neck region or regions necessitating overlapping fields
3. Concurrent use of any anti- cancer treatment, standard, alternative or investigational.
4. History of allergic reactions to any agents in this study
5. Autoimmune disease or organ transplant which in the judgment of the PI would increase the risk of immune checkpoint inhibition.
6. Pregnant or breastfeeding
7. Severe, active co-morbidity, defined as follows:

   * Major medical or psychiatric illness, which in the investigator's opinion would interfere with the completion of therapy and follow up or with full understanding of the risks and potential complications of the therapy;
   * Unstable angina and/or uncontrolled congestive heart failure within past 6 months;
   * Myocardial infarction within the last 6 months;
   * Current acute bacterial or fungal infection requiring intravenous antibiotics; note that patients receiving IV antibiotics or currently on oral antibiotics whose infection is assessed to be adequately treated or controlled are eligible.
   * Chronic Obstructive Pulmonary Disease exacerbation or other respiratory illness requiring hospitalization or precluding study therapy within 30 days prior to day 1 of treatment;
8. Acquired Immune Deficiency Syndrome (AIDS) based upon current CDC definition; note, however, that HIV testing is not required for entry into this protocol. The need to exclude patients with AIDS from this protocol is necessary because the treatments involved in this protocol may be significantly immunosuppressive
9. Patients with hearing loss assessed to be primarily sensorineural in nature, requiring a hearing aid, or intervention (i.e. interfering in a clinically significant way with activities of daily living); a conductive hearing loss that is tumor-related is allowed
10. ≥ grade 2 peripheral sensory neuropathy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2024-09-03 (Actual); Primary Completion 2029-01 (Estimated); Study Completion 2029-01 (Estimated)

PRIMARY OUTCOMES:
Induction chemotherapy completion rate | 3 years
  Induction chemotherapy completion rate, defined as the proportion of patients who complete three cycles of chemoimmunotherapy within 12 weeks of initiation. Completion is defined for induction as receiving all 3 cycles as planned, including protocol specified dose reduction and delays. .
Radiation completion rate | 3 years
  Radiation completion rate, defined as the proportion of patients who complete specified radiation within 8 weeks of radiation initiation. Radiation completion is defined as completion of planned doses of radiation.

SECONDARY OUTCOMES:
Overall Response (ORD) rate following induction | 3 years
  OR rate following induction, defined as the proportion of patients who achieve at least a RECIST defined PR within 12 weeks of induction chemotherapy initiation.
Complete Response (CR) rate following radiation | 3 years
  CR rate following radiation, defined as the proportion of patients who achieve a RECIST defined CR within 16 weeks following the end of radiation therapy.

CONTACTS AND LOCATIONS:
Overall Officials: A. Dimitrios Colevas, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford University, Palo Alto, California, United States